CLINICAL TRIAL: NCT04443946
Title: Different Anesthesia Maintain Protocol Effect the Outcome of the Patients Undergoing General Anesthesia for Urinary Surgery
Brief Title: Different Anesthesia Maintain Protocol Effect the Outcome of the Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CINI-AD-20205-19
Record Dates: First submitted 2020-06-08; First posted 2020-06-23 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-06

CONDITIONS: Urinary Surgery; General Anesthesia
MeSH Terms: interventions — Propofol; Sevoflurane; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group-P (Active Comparator): Group-P: (Propofol group): 5 mg kg-1 h-1 propofol was pumped continuously after endotracheal intubation.
  Interventions: Drug: Propofol
- Group-PAS (Experimental): Group-PAS: (Propofol and after 20 min adding Sevoflurane group): 2.5 mg kg-1 h-1 propofol were pumped continuously and add 1% end-tidal sevoflurane 20 minutes after endotracheal intubation.
  Interventions: Drug: 1% Sevoflurane; Drug: Propofol half
- Group-PS (Experimental): Group-PS: (Propofol and Sevoflurane group): 2.5 mg kg-1 h-1 propofol were continuously pumped after endotracheal intubation, and 1% sevoflurane was inhaled continuously at the same time.
  Interventions: Drug: 1% Sevoflurane continue; Drug: Propofol half
- Group-S (Experimental): Group-S: (Sevoflurane group): 2% sevoflurane continued to maintain anesthesia after endotracheal intubation.
  Interventions: Drug: 2% Sevoflurane
- Group-PSu (Experimental): Group-PSu: (Propofol and Sufentanil group): 5 mg kg-1 h-1 propofol, 0.01 μ g kg-1 min-1 sufentanil were pumped continuously at maintain phase
  Interventions: Drug: Propofol; Drug: Sufentanil

INTERVENTIONS:
Drug: Propofol — 5 mg kg-1 h-1 propofol was pumped continuously after endotracheal intubation.
  Arms: Group-P; Group-PSu
Drug: 1% Sevoflurane — add 1% end-tidal sevoflurane 20 minutes after endotracheal intubation.
  Arms: Group-PAS
Drug: 1% Sevoflurane continue — 1% sevoflurane continued to maintain anesthesia after endotracheal intubation.
  Other Names: 1% Sevoflurane
  Arms: Group-PS
Drug: Sufentanil — 0.01 μ g kg-1 min-1 sufentanil were pumped continuously at maintain phase
  Arms: Group-PSu
Drug: 2% Sevoflurane — 2% sevoflurane continued to maintain anesthesia after endotracheal intubation.
  Other Names: 2% Sevoflurane continue
  Arms: Group-S
Drug: Propofol half — 2.5 mg kg-1 h-1 propofol was pumped continuously after endotracheal intubation.
  Other Names: 2.5% Propofol
  Arms: Group-PAS; Group-PS

SUMMARY:
This prospective open-label randomized study, patients were having elective urological surgery scheduled to last longer than 1 h under necessitating general anesthesia.Group-P: (Propofol group): 3 mg kg-1 min-1 propofol was pumped continuously after endotracheal intubation. Group-PAS: (Propofol and after 20 min adding Sevoflurane group): 3 mg kg-1 min-1 propofol were pumped continuously and add 1% end-tidal sevoflurane 20 minutes after endotracheal intubation. Group-PS: (Propofol and Sevoflurane group): 3 mg kg-1 min-1 propofol were continuously pumped after endotracheal intubation, and 1% sevoflurane was inhaled continuously at the same time. Group-S: (Sevoflurane group): 1% sevoflurane continued to maintain anesthesia after endotracheal intubation. Group-PSu: (Propofol and Sufentanil group): 3 mg kg-1 min-1 propofol, 0.01 μ g kg-1 min-1 sufentanil were pumped continuously at maintain phase

DETAILED DESCRIPTION:
Group-P: (Propofol group): 3 mg kg-1 min-1 propofol was pumped continuously after endotracheal intubation. Group-PAS: (Propofol and after 20 min adding Sevoflurane group): 3 mg kg-1 min-1 propofol were pumped continuously and add 1% end-tidal sevoflurane 20 minutes after endotracheal intubation. Group-PS: (Propofol and Sevoflurane group): 3 mg kg-1 min-1 propofol were continuously pumped after endotracheal intubation, and 1% sevoflurane was inhaled continuously at the same time. Group-S: (Sevoflurane group): 1% sevoflurane continued to maintain anesthesia after endotracheal intubation. Group-PSu: (Propofol and Sufentanil group): 3 mg kg-1 min-1 propofol, 0.01 μ g kg-1 min-1 sufentanil were pumped continuously at maintain phase. Due to the ethical requirements of adequent analgesia, 0.3 μ g kg-1 min-1 remifentanil was continuously pumped as background input dose during anesthesia maintenance in all groups.

ELIGIBILITY:
Inclusion Criteria:

* the aged 18-65 yr,
* ASA physical status I, II or III patients
* having elective urological surgery
* operation scheduled to last longer than 1 h
* under necessitating general anesthesia

Exclusion Criteria:

* refused to participate in the study;
* were not able to communicate due to alterations in the level of consciousness, - a history of allergy to opioids
* contraindications inhalational anaesthesia
* family history of malignant hyperthermia
* alcohol or drug abuse
* received central nervous system-active drugs;
* body mass index ≥40 kg/m2
* represent conditions liable to alter the pharmacokinetic and pharmacodynamic behaviors of the intravenous and inhalation anesthetics
* previous head injury, neurologic or psychiatric disease
* any disabling central nervous
* cerebrovascular disease
* current use of psychoactive or anti-convulsive medications
* unstable angina
* manifest congestive heart failure
* airway management was expected to be difficult

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Extubation Duration(ED) | Up to 24 hours
  the extubation Duration (ED) was calculated as the time from the end of anesthesia to extubation of the LMA

SECONDARY OUTCOMES:
Length of PACU | Up to 24 hours
  Length of PACU (Post-anesthesia care unit): From entering the PACU to discharge from the PACU
qNOX | From entering the operation room until the discharge from the operation room, assessed up to 12 hours
  Noceciption index,The qNOX of depth of analgesia also ranges from 99 to 0, and usually it is controlled to be within 40-60 during the operative period, with qNOX > 80 indicating an insufficient use of analgesic agents and qNOX < 10 indicating excessive analgesic effects.
Bis | From entering the operation room until the discharge from the operation room, assessed up to 12 hours
  Bispectral index,Bis 50-80 means appropriate Sedation depth
Blood pressure | From entering the operation room until the discharge from the operation room, assessed up to 12 hours
  measuring Systolic, Diastolic and Mean Blood Pressure
The heart rate | From entering the operation room until the discharge from the operation room, assessed up to 12 hours
  The heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Yanghai Cui, Study Chair — China International Neuroscience Institution
Locations (1):
- Xuanwu hospital, Beijing, Beijing Municipality, China